CLINICAL TRIAL: NCT01712555
Title: Autologous Fat Grafting to Anophthalmic Sockets With PRP (Platelet Rich Plasma) Using a Closed Cannula Technique
Brief Title: Autologous Fat Grafting With PRP (Platelet Rich Plasma) to Anophthalmic Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox, Donald Munro, M.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: New York Eye and Ear Infirmary
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Orbital Atrophy
Keywords: Anophthalmic orbits; autologous fat; platelet rich plasma; orbital atrophy; anophthalmos; cannula
MeSH Terms: conditions — Anophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fat grafting with PRP to anophthalmic orbits (Experimental): There is only one arm to this study. People with orbital atrophy and loss of an eye are to be injected with autologous fat mixed with autologous PRP (platelet rich plasma) and observed for at least one year for evidence of retention of the injected fat
  Interventions: Procedure: autologous fat grafting with PRP to anophthalmic orbits

INTERVENTIONS:
Procedure: autologous fat grafting with PRP to anophthalmic orbits

SUMMARY:
After people lose an eye, for whatever reason, they often experience fat atrophy of the tissues in the orbit. This leads to a sunken appearance that is often not correctable by a cosmetic shell prosthesis. Current techniques to correct this deformity are inadequate/ invasive. Injection of various gels (Restylane, Radiesse) are temporary had have their own disadvantages. This study seeks to demonstrate an improvement in the retention of injected autologous fat by mixing in autologous PRP (platelet rich plasma).

ELIGIBILITY:
Inclusion Criteria: anophthalmos, orbital atrophy -

Exclusion Criteria:poor anesthesia risk, people outside a 100 mile radius of New York City

-

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Improved retention of autologous fat injected into anophthalmic sockets | 1-5 yrs
  Non contrast MRIs of the orbits are obtained before, immediately after, and one year after injection of autologous fat mixed with autologous PRP (platelet rich plasma)

CONTACTS AND LOCATIONS:
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States

REFERENCES:
- See also: related info — http://www.newyorkfami.com